CLINICAL TRIAL: NCT04714931
Title: Sentinel Lymph Node Assessment In Ovarian Cancer - Turkish Gynecologic Oncology Group Study (TRSGO-SLN-005)
Brief Title: Sentinel Lymph Node Assessment in Ovarian Cancer (TRSGO-SLN-OO5)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Ozguc Takmaz, MD,Assistant Professor, Acibadem University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TRSGO-SLN-OO5
Record Dates: First submitted 2021-01-13; First posted 2021-01-20 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Ovarian Cancer; Sentinel Lymph Node
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective, Controlled, not randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sentinel Lymph Node (Other): Sentinel lymph nodes which can be identified with the tracer involvement will be removed. Then, systematic lymphadenectomy will be performed according to the routine practice.
  Interventions: Diagnostic Test: Sentinel lymph node detection

INTERVENTIONS:
Diagnostic Test: Sentinel lymph node detection — Tracer (Indocyanine green or blue dye) will be injected into the IP and utero-ovarian ligaments, after opening of the pelvic and paraaortic retroperitoneal spaces, sentinel lymph nodes which can be identified with the tracer involvement will be removed. Then, systematic lymphadenectomy will be performed according to the routine practice.

SUMMARY:
The aim of the study to evaluate the feasibility and accuracy of sentinel lymph node technique in ovarian cancer.

DETAILED DESCRIPTION:
Systematic pelvic and paraaortic lymphadenectomy is commonly performed in ovarian cancer patients. However, in early ovarian cancer systematic lymphadenectomy can be an unnecessary procedure which can cause perioperative morbidity and mortality. In the other hand, initially diagnosed early stage ovarian cancer can be upstaged after staging surgery with systematic lymphadenectomy. For preventing unnecessary lymphadenectomy in early ovarian cancer, sentinel lymph node procedure may be an alternative which can prevent major complications without missing the real stage of the disease.

Aim of our study is to assess the feasibility and accuracy of lymph node evaluation with sentinel lymph node technique in early ovarian cancer patients. Pelvic and paraaortic spaces will be evaluated for the sentinel lymph nodes after the injection of the tracers in infundibulopelvic and utero-ovarian ligaments. Than routine systematic pelvic and paraaortic lymphadenectomy will be performed with the routine practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Early stage ovarian cancer

Exclusion Criteria:

* Patient who had been administrated chemotherapy prior to surgery
* Patients who had diagnosed with malignancy other than ovarian cancer.
* Patients who had undergone pelvic or paraaortic lymphadenectomy or surgery prior to surgery.
* Patients who have allergy for the tracers.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Sentinel lymph node localization | 12 months
  Localization areas of pelvic and paraaortic sentinel lymph nodes for ovarian cancer will be identified.
Sentinel lymph node technique accuracy in ovarian cancer | 12 months
  Sensitivity and specificity measure of the sentinel lymph node procedure in ovarian cancer for detecting the lymphatic metastasis
PPV and NPV of sentinel lymph node procedure in ovarian cancer | 12 months
  Positive predictive and negative predictive value of sentinel lymph node procedure in ovarian cancer.
Adverse events | 12 months
  Adverse events related with sentinel lymph node procedure in ovarian cancer
Sentinel lymph node detection rate | 12 months
  Pelvic and paraaortic Sentinel lymph node detection rates will be assessed for ovarian cancer.

SECONDARY OUTCOMES:
Tracer comparisons | 12 months
  Detection rate differences between different tracers
Assessment of the sentinel tecniques | 12 months
  Evaluation of the tracer injection techniques whether before the excision of the mass or after the excision of the mass for the effectiveness of sentinel lymph node detection.

CONTACTS AND LOCATIONS:
Overall Officials: Mete Gungor, Prof., Study Director — Acibadem MAA University Maslak Hospital
Locations (1):
- Acibadem MAA University Maslak Hospital, Istanbul, Turkey (Türkiye)